CLINICAL TRIAL: NCT03066375
Title: Diagnostic Accuracy of the Inferior Vena Cava Collapsibility to Predict Fluid Responsiveness in Spontaneously Breathing Patients With Sepsis, Acute Circulatory Failure, and Irregular Cardiac Rhythm
Brief Title: Respiratory Variations For Predicting Fluid Responsiveness 2
Acronym: ReVaPreF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011_46; 2011-A01598-33 (Other: ID-RCB number)
Record Dates: First submitted 2016-11-09; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Sepsis; Circulatory Failure; Respiratory Physiological Phenomena
Keywords: vena cava; fluid; sepsis; echocardiography; ultrasound; ultrasonography; collapsibility index; circulatory failure; irregular cardiac rhythm; fluid responsiveness; Spontaneous breathing
MeSH Terms: conditions — Sepsis; Shock | interventions — Echocardiography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echocardiography-Doppler (Experimental): Ultrasonographic recordings, systemic arterial pressure, heart rate, and respiratory rate are recorded immediately before and after volume expansion (VE), performed as a 30-minute infusion of 500 mL of 4% gelatin. Inferior Vena Cava diameters are measured during spontaneous and standardized respiratory cycles. Stroke volume is measured during spontaneous respiratory cycles.
  Interventions: Device: Echocardiography-Doppler

INTERVENTIONS:
Device: Echocardiography-Doppler — Ultrasonographic recordings are recorded immediately before and after volume expansion (VE), performed as a 30-minute infusion of 500 mL of 4% gelatin. Inferior Vena Cava diameters are measured during spontaneous and standardized respiratory cycles. Stroke volume is measured during spontaneous respiratory cycles.

SUMMARY:
Objectives: To investigate whether respiratory variations of inferior vena cava diameters (cIVC) predict fluid responsiveness in spontaneously breathing patients with septic acute circulatory failure and irregular heartbeats.

Design: Prospective, bicentric study, intensive care units.

Patients and measures: Spontaneously breathing patients with sepsis and clinical signs of acute circulatory failure are included. A positive response to fluid loading (FL) is defined as an increase of the stroke volume (SV) >10%. The investigators measured the minimum inspiratory and maximum expiratory diameters of the IVC (idIVC and edIVC) during standardized (st) and unstandardized (ns) breathing. The investigators calculated cIVCst and cIVCns before a 500ml-colloid FL.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of the intensive care units of the Lille university-hospital and of the Valencienne general hospital.
* Age greater than or equal to 18.
* Patient insured
* Spontaneous breathing without ventilatory support or intubation or tracheotomy.
* Irregular cardiac rhythm
* Prescription by the physician in charge of the patients of a 500 mL volume expansion in less than 30 minutes.
* Patients with sepsis with at least one sign of acute circulatory failure:

  * Tachycardia with heart rate> 100/min
  * systolic blood pressure <90mmHg or a decrease >40mmHg in previously hypertense patient
  * Oliguria <0.5ml/kg/hour for at least one hour
  * skin mottling

Exclusion Criteria:

* high-grade aortic insufficiency
* transthoracic echogenicity unsuitable for measuring the stroke volume or inferior vena cava diameters
* clinical signs of active exhalation
* clinical or ultrasonographic evidence of pulmonary edema due to heart failure
* pregnancy
* abdominal compartment syndrome
* regular cardiac rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
respiratory variations in inferior vena cava diameters with respect to the response to fluid resuscitation, assessed by the area under the ROC curve | during 30 minutes of the volume expansion

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Preau, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Intensive Care Department, Salengro Hospital,CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No